CLINICAL TRIAL: NCT04429412
Title: Effectiveness of the Individualized Metacognitive Training (EMC+) in People With Psychosis of Brief Evolution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: Parc Sanitari Sant Joan de Déu (Other); Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other); Servicio Andaluz Jaén y Málaga (Unknown); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); Parc de Salut Mar (Other); Centre d'Higiene Mental Les Corts (Other); Institut Pere Mata (Unknown); Institut Assistència Sanitària Girona (Unknown); Hospital Clínico Universitario de Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI14/00044
Record Dates: First submitted 2020-06-01; First posted 2020-06-12 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-05

CONDITIONS: Brief Psychotic Disorder; Psychosis; Episode
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: This is a randomized clinical trial in which some patients receive the EMC+ and others treatment as usual.
Who Masked: Outcomes Assessor
Masking Description: The evaluator will be blind to the group that owns the patients included.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metacognitive Training (MCT+) (Experimental): MCT+ combines the process-oriented approach of metacognitive group training with elements of individual cognitive-behavioral therapy.
  The metacognitive training program is comprised of 10 modules targeting common cognitive errors in schizophrenia. (Moritz et al, 2013).
  The modules are: 1:Therapeutic alliance, 2: Introducyion to MCT+, 3:Disease model, 4: Attributional style, 5: Decision making, 6: Changing beliefs, 7: Empathizing, 8: Memory, 9: Depression and self-steem, 10: Relapse prevention.
  The treatment consist of 10 weekly sessions of 45-60 minutes.
  Interventions: Behavioral: MCT+
- TAU (No Intervention): Treatment as usual.

INTERVENTIONS:
Behavioral: MCT+ — Metacognitive training
  Arms: Metacognitive Training (MCT+)

SUMMARY:
The main aim of the study is to evaluate the effectiveness of Individualized Meta-Cognitive Training (EMC +), in people with psychosis of brief evolution on symptoms, especially on positive symptoms. Secondary aims would be to assess the effect of EMC+ in metacognition, psychosocial and neuropsychological functioning, and to assess the maintenance of program effects on 6 months.

DETAILED DESCRIPTION:
This is a randomized clinical trial in which some patients receive the EMC+ and others treatment as usual.The evaluator will be blind to the group to which the patients belong. The sample for the overall project will be a total of 70 people with a diagnosis of psychotic spectrum, less than 5 years of experience and with a score => 3 positive PANSS (last month) and treated in one of the participating institutions. The evaluation was performed at baseline, at post-treatment and at 6 months follow up. Symptoms, metacognition, psychosocial and neuropsychological functioning were assessed.

The EMC consists of 10 therapeutic units with weekly sessions of 45-60 minutes. The material available for the Individualized Metacognitive Training (EMC) program is made up of power-point presentations.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of : schizophrenia, schizoaffective disorder, brief psychotic disorder, delusional disorder, schizophreniform disorder, psychotic disorder not otherwise specified.
* Less than 5 years of evolution.
* Score at or above 4 on the PANSS during the last year (delusions, grandiosity, suspiciousness).

Exclusion Criteria:

* Traumatic brain injury, dementia, or intellectual disability (premorbid IQ ≤70).
* Substance dependence.
* Score at or above 5 on the PANSS ( Hostility and Uncooperativeness); score at or above 6 on the PANSS (suspiciousness).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
PANSS. Positive and Negative Syndrome Scale. (Kay et al., 1987; Peralta and Cuesta, 1994) | baseline.
  The Positive and Negative Syndrome Scale (PANSS). This scale measures 30 symptoms on a scale of 1-7, with higher scores indicating greater psychopathology. The PANSS contains three sub-scales: positive, negative and general symptoms. Range: 7-112. Higher values represent a worse outcome.
PANSS. Positive and Negative Syndrome Scale. (Kay et al., 1987; Peralta and Cuesta, 1994) | immediately after the intervention
  The Positive and Negative Syndrome Scale (PANSS). This scale measures 30 symptoms on a scale of 1-7, with higher scores indicating greater psychopathology. The PANSS contains three sub-scales: positive, negative and general symptoms.Range: 7-112. Higher values represent a worse outcome.
PANSS. Positive and Negative Syndrome Scale. (Kay et al., 1987; Peralta and Cuesta, 1994) | 6 months follow-up
  The Positive and Negative Syndrome Scale (PANSS). This scale measures 30 symptoms on a scale of 1-7, with higher scores indicating greater psychopathology. The PANSS contains three sub-scales: positive, negative and general symptoms.Range: 7-112. Higher values represent a worse outcome.

SECONDARY OUTCOMES:
Jumping to conclusions. (Brett-Jones et al. 1987). | baseline
  Three different computer tasks were used in the study. In Task 1, jars contained balls of two different colors; in one of them the proportion was 85 black versus 15 orange balls and in the other the ratio was reversed. Task 2 was the same as Task 1 but with a proportion of 60:40 in each jar. Finally, Task 3 was similar to Task 2 but instead of balls, the jars contained positive or negative comments with a proportion of 60:40. The patients had to decide which to jar belonged the extracted balls or comments. At all times the participants had information about the balls previously extracted, in order to control the effect of memory. The subjects could remove as many balls as needed to make their final decision (Garety et al., 2005). JTC was considered as taking a decision after extracting 1 or 2 balls.Dichotomous: yes/no. A "yes" represents a worse outcome
Jumping to conclusions. (Brett-Jones et al. 1987). | immediately after the intervention
  Three different computer tasks were used in the study. In Task 1, jars contained balls of two different colors; in one of them the proportion was 85 black versus 15 orange balls and in the other the ratio was reversed. Task 2 was the same as Task 1 but with a proportion of 60:40 in each jar. Finally, Task 3 was similar to Task 2 but instead of balls, the jars contained positive or negative comments with a proportion of 60:40. The patients had to decide which to jar belonged the extracted balls or comments. At all times the participants had information about the balls previously extracted, in order to control the effect of memory. The subjects could remove as many balls as needed to make their final decision (Garety et al., 2005). JTC was considered as taking a decision after extracting 1 or 2 balls.Dichotomous: yes/no. A "yes" represents a worse outcome
Jumping to conclusions. (Brett-Jones et al. 1987). | 6 months follow-up
  Three different computer tasks were used in the study. In Task 1, jars contained balls of two different colors; in one of them the proportion was 85 black versus 15 orange balls and in the other the ratio was reversed. Task 2 was the same as Task 1 but with a proportion of 60:40 in each jar. Finally, Task 3 was similar to Task 2 but instead of balls, the jars contained positive or negative comments with a proportion of 60:40. The patients had to decide which to jar belonged the extracted balls or comments. At all times the participants had information about the balls previously extracted, in order to control the effect of memory. The subjects could remove as many balls as needed to make their final decision (Garety et al., 2005). JTC was considered as taking a decision after extracting 1 or 2 balls.Dichotomous: yes/no. A "yes" represents a worse outcome
BCIS. Beck Cognitive and Insight Scale. (Beck et al., 2004; Gutierrez-Zotes et al., 2012) | baseline
  The Beck Cognitive Insight Scale. this scale is a self-registering measure of 15 items .which evaluates how the patients assess their own judgement. It has two dimensions; self-reflection (R) (9 items), and self-certainty (C) (6 items). A compound index of cognitive insight is obtained as the subtraction of self-certainty from self-reflection (R-C).Range: 0-45. Higher values represent a better outcome
BCIS. Beck Cognitive and Insight Scale. (Beck et al., 2004; Gutierrez-Zotes et al., 2012) | immediately after the intervention
  The Beck Cognitive Insight Scale. this scale is a self-registering measure of 15 items .which evaluates how the patients assess their own judgement. It has two dimensions; self-reflection (R) (9 items), and self-certainty (C) (6 items). A compound index of cognitive insight is obtained as the subtraction of self-certainty from self-reflection (R-C).Range: 0-45. Higher values represent a better outcome
BCIS. Beck Cognitive and Insight Scale. (Beck et al., 2004; Gutierrez-Zotes et al., 2012) | 6 months follow-up
  The Beck Cognitive Insight Scale. this scale is a self-registering measure of 15 items .which evaluates how the patients assess their own judgement. It has two dimensions; self-reflection (R) (9 items), and self-certainty (C) (6 items). A compound index of cognitive insight is obtained as the subtraction of self-certainty from self-reflection (R-C).Range: 0-45. Higher values represent a better outcome
IPSAQ. Internal, Personal and Situational Attribution Questionnaire. (Kinderman & Bentall, 1996) | baseline
  The scale assess the attributional style in 32 situations. Personalizing Bias (PB) indicates the proportion of external attributions for negative events which are personal as opposed to situational. A PB score of greater than 0.5 therefore represents a greater tendency to use personal rather than situational external attributions for negative events.
IPSAQ. Internal, Personal and Situational Attribution Questionnaire. (Kinderman & Bentall, 1996) | immediately after the intervention
  The scale assess the attributional style in 32 situations. Personalizing Bias (PB) indicates the proportion of external attributions for negative events which are personal as opposed to situational. A PB score of greater than 0.5 therefore represents a greater tendency to use personal rather than situational external attributions for negative events.
IPSAQ. Internal, Personal and Situational Attribution Questionnaire. (Kinderman & Bentall, 1996) | 6 months follow-up
  The scale assess the attributional style in 32 situations. Personalizing Bias (PB) indicates the proportion of external attributions for negative events which are personal as opposed to situational. A PB score of greater than 0.5 therefore represents a greater tendency to use personal rather than situational external attributions for negative events.
The Hinting Task. (Corcoran et al. 1995; Gil et al. 2012) | baseline
  The Scale assess Theory of Mind.Possible range: 0-12. Higher values represent a better outcome
The Hinting Task. (Corcoran et al. 1995; Gil et al. 2012) | immediately after the intervention
  The Scale assess Theory of Mind. Possible range: 0-12. Higher values represent a better outcome
The Hinting Task. (Corcoran et al. 1995; Gil et al. 2012) | 6 months follow-up
  The Scale assess Theory of Mind. Possible range: 0-12. Higher values represent a better outcome
Emotional Recognition Test Faces. (Baron-Cohen et al. 1997) | baseline
  20 photographs that express ten basic and ten complex emotions.Possible range: 0-20. Higher values represent a better outcome
Emotional Recognition Test Faces. (Baron-Cohen et al. 1997) | immediately after the intervention
  20 photographs that express ten basic and ten complex emotions. Possible range: 0-20. Higher values represent a better outcome
Emotional Recognition Test Faces. (Baron-Cohen et al. 1997) | 6 months follow-up
  20 photographs that express ten basic and ten complex emotions.Possible range: 0-20. Higher values represent a better outcome
MASC. (Lahera et al.2014). | immediately after the intervention
  A Movie for the Assessment of Social Cognition. Spanish Validation. 46 multiple-choice questions about the emotions, thoughts or intentions of the protagonists.
  Only one answer out of four is correct. The four choices of each answer include, (1) correct attribution of ToM to the characters of the film, (2) excessive ToM errors (a mental state that is attributed when there is no reason to), (3) reduced ToM errors (a present mental state that is not attributed) and (4) total absence of mental inference (a physical causality attribution instead of a mental state). These errors could be classified as overmentalization, undermentalization and absence of mentalization.

OTHER OUTCOMES:
SFS. Social Functioning Scale.(Birchwood et al, 1990; Torres y Olivares, 2000). | baseline
  This scale assess social functioning in people with psychotic disorders. Range: 45-195
SFS. Social Functioning Scale.(Birchwood et al, 1990; Torres y Olivares, 2000). | immediately after the intervention
  This scale assess social functioning in people with psychotic disorders.Range: 45-195
SFS. Social Functioning Scale.(Birchwood et al, 1990; Torres y Olivares, 2000). | 6 months follow-up
  This scale assess social functioning in people with psychotic disorders.Range: 45-195
WCST(Wisconsin Card Sorting Test, Bergs et al, 1948) | baseline
  measure of executive function. Categories completed and perseverative errors. Higher values represent a better outcome.
WCST(Wisconsin Card Sorting Test, Bergs et al, 1948) | immediately after the intervention
  measure of executive function. Categories completed and perseverative errors. Higher values represent a better outcome.
WCST(Wisconsin Card Sorting Test, Bergs et al, 1948) | 6 months follow-up
  measure of executive function. Categories completed and perseverative errors. Higher values represent a better outcome.
Test Stroop (Stroop, 1935) | baseline
  flexibility and inhibition of automatic responses.Higher values represent a better outcome.
Test Stroop (Stroop, 1935) | immediately after the intervention
  flexibility and inhibition of automatic responses.Higher values represent a better outcome.
Test Stroop (Stroop, 1935) | 6 months follow-up
  flexibility and inhibition of automatic responses.Higher values represent a better outcome.
TMT A B (Trail Making Test, Reitan, 1993) | baseline
  visual attention and task switching. Higher values represent a worse outcome.
TMT A B (Trail Making Test, Reitan, 1993) | immediately after the intervention
  visual attention and task switching. Higher values represent a worse outcome.
TMT A B (Trail Making Test, Reitan, 1993) | 6 months follow-up
  visual attention and task switching. Higher values represent a worse outcome.
CPT-IP (Continous Performance Test, Matrics) | baseline
  measure of attention. Higher values represent a better outcome.
CPT-IP (Continous Performance Test, Matrics) | 6 months follow-up
  measure of attention.Higher values represent a better outcome.
TAVEC (Verbal Learning Test), Benedet and Aleixandre 1998) | baseline
  measure of verbal memory.Higher values represent a better outcome.
TAVEC (Verbal Learning Test), Benedet and Aleixandre 1998) | 6 months follow-up
  measure of verbal memory. Higher values represent a better outcome.
WAIS-III (Weschler Adults Intelligence Scale, Wechsler 1955) | baseline
  vocabulary subscale. Higher values represent a better outcome.
WAIS-III (Weschler Adults Intelligence Scale, Wechsler 1955) | baseline
  digits subscale. Higher values represent a better outcome.
WAIS-III (Weschler Adults Intelligence Scale, Wechsler 1955) | immediately after the intervention
  digits subscale. Higher values represent a better outcome.
WAIS-III (Weschler Adults Intelligence Scale, Wechsler 1955) | 6 months follow-up
  digits subscale. Higher values represent a better outcome.